CLINICAL TRIAL: NCT03242252
Title: A Randomized, Double-blind, Placebo-controlled, 3-arm, Parallel-group 52-week Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin in Patients With Type 2 Diabetes Mellitus and Moderate Renal Impairment Who Have Inadequate Glycemic Control
Brief Title: Safety and Efficacy Study of Sotagliflozin on Glucose Control in Participants With Type 2 Diabetes, Moderate Impairment of Kidney Function, and Inadequate Blood Sugar Control
Acronym: SOTA-CKD3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC14837; 2016-004889-26; U1111-1187-8662 (Other: UTN)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease Stage 3
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Following a 2-week run-in period, participants received two placebo tablets (identical to sotagliflozin 200 mg in appearance), orally once daily, before the first meal of the day for up to 54 weeks.
  Interventions: Drug: Placebo
- Sotagliflozin 200 mg (Experimental): Following a 2-week run-in period, participants received two tablets, 1 sotagliflozin 200 mg tablet and 1 placebo tablet (identical to sotagliflozin 200 mg in appearance), orally once daily, before the first meal of the day for up to 58 weeks.
  Interventions: Drug: Placebo; Drug: Sotagliflozin
- Sotagliflozin 400 mg (Experimental): Following a 2-week run-in period, participants received sotagliflozin 400 mg, administered as two 200 mg sotagliflozin tablets, orally once daily, before the first meal of the day for up to 60 weeks.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Placebo — Placebo tablet (identical to sotagliflozin 200 mg in appearance), orally once daily.
  Route of administration: Oral
  Arms: Placebo; Sotagliflozin 200 mg
Drug: Sotagliflozin — Sotagliflozin 200 mg, tablet, orally once daily.
  Route of administration: Oral
  Other Names: SAR439954
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg

SUMMARY:
Primary Objective:

To demonstrate the superiority of Sotagliflozin 200 milligrams (mg) and Sotagliflozin 400 mg versus placebo on HbA1c reduction at 26 Weeks in participants with Type 2 diabetes who have inadequate glycemic control and moderate renal impairment.

Secondary Objectives:

* To assess the effects of Sotagliflozin 200 mg and 400 mg versus placebo with respect to additional measures of glycemic control, blood pressure, and body weight.
* To evaluate the safety of Sotagliflozin 200 mg and 400 mg versus placebo.

DETAILED DESCRIPTION:
The study duration is up to 60 weeks including 4 weeks prior to randomization, 52 weeks of randomized treatment, and a visit 4 weeks after completion of the randomized treatment period.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 Diabetes (drug-naïve or on antidiabetic therapy) and documented moderate renal insufficiency defined by an estimated glomerular filtration rate (eGFR) (based on the 4 variable Modification of Diet in Renal Disease (MDRD) equation) of ≥30 and <60 milliliter per minute (mL/min)/1.73 meter square (m^2) (chronic kidney disease [CKD] 3A, 3B).
* Participants has given written informed consent to participate in the study in accordance with local regulations.

Exclusion criteria:

* Hemoglobin A1c (HbA1c) of <7.0% or >11.0%.
* Type 1 diabetes.
* Women of childbearing potential (WOCBP) not willing to use highly effective method(s) of birth control during the study treatment period and the follow-up period, or who are unwilling or unable to be tested for pregnancy during the study.
* Treatment with a sodium-glucose cotransporter type 2 (SGLT2) inhibitor (Canagliflozin, Dapagliflozin, Empagliflozin) during the last 12 months.
* Uncontrolled high blood pressure.
* Participants with severe anemia, severe cardiovascular (including congestive heart failure New York Heart Association IV), respiratory, hepatic, neurological, psychiatric, or active malignant tumor or other major systemic disease or patients with short life expectancy that, according to the Investigator, will preclude their safe participation in this study, or will make implementation of the protocol or interpretation of the study results difficult.
* Lower extremity complications (such as skin ulcers, infection, osteomyelitis and gangrene) identified during the Screening period, and still requiring treatment at Randomization.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (170):
- United States (51):
  - Investigational Site Number 8404018, Birmingham, Alabama
  - Investigational Site Number 8404045, Guntersville, Alabama
  - Investigational Site Number 8404004, Phoenix, Arizona
  - Investigational Site Number 8404022, Phoenix, Arizona
  - Investigational Site Number 8404007, Little Rock, Arkansas
  - Investigational Site Number 8404023, Chula Vista, California
  - Investigational Site Number 8404044, Gold River, California
  - Investigational Site Number 8404011, Los Angeles, California
  - Investigational Site Number 8404003, Norco, California
  - Investigational Site Number 8404025, Northridge, California
  - Investigational Site Number 8404038, San Dimas, California
  - Investigational Site Number 8404019, Clearwater, Florida
  - Investigational Site Number 8404001, DeLand, Florida
  - Investigational Site Number 8404006, Ocoee, Florida
  - Investigational Site Number 8404064, Orlando, Florida
  - Investigational Site Number 8404043, Ormond Beach, Florida
  - Investigational Site Number 8404013, Palmetto Bay, Florida
  - Investigational Site Number 8404016, Savannah, Georgia
  - Investigational Site Number 8404040, Wauconda, Illinois
  - Investigational Site Number 8404036, Lake Charles, Louisiana
  - Investigational Site Number 8404020, New Orleans, Louisiana
  - Investigational Site Number 8404014, Norfolk, Nebraska
  - Investigational Site Number 8404032, Papillion, Nebraska
  - Investigational Site Number 8404048, Hackensack, New Jersey
  - Investigational Site Number 8404074, New York, New York
  - Investigational Site Number 8404009, The Bronx, New York
  - Investigational Site Number 8404051, Wilmington, North Carolina
  - Investigational Site Number 8404028, Winston-Salem, North Carolina
  - Investigational Site Number 8404029, Winston-Salem, North Carolina
  - Investigational Site Number 8404026, Dayton, Ohio
  - Investigational Site Number 8404052, Lansdale, Pennsylvania
  - Investigational Site Number 8404031, Anderson, South Carolina
  - Investigational Site Number 8404021, Mt. Pleasant, South Carolina
  - Investigational Site Number 8404056, Chattanooga, Tennessee
  - Investigational Site Number 8404015, Austin, Texas
  - Investigational Site Number 8404050, Austin, Texas
  - Investigational Site Number 8404060, Austin, Texas
  - Investigational Site Number 8404005, Beaumont, Texas
  - Investigational Site Number 8404035, Dallas, Texas
  - Investigational Site Number 8404039, Houston, Texas
  - Investigational Site Number 8404055, Houston, Texas
  - Investigational Site Number 8404012, Hurst, Texas
  - Investigational Site Number 8404033, Lampasas, Texas
  - Investigational Site Number 8404053, McAllen, Texas
  - Investigational Site Number 8404057, Round Rock, Texas
  - Investigational Site Number 8404059, San Antonio, Texas
  - Investigational Site Number 8404010, San Antonio, Texas
  - Investigational Site Number 8404008, Layton, Utah
  - Investigational Site Number 8404042, Renton, Washington
  - Investigational Site Number 8404041, Seattle, Washington
  - Investigational Site Number 8404047, Kenosha, Wisconsin
- Argentina (7):
  - Investigational Site Number 0324001, Buenos Aires
  - Investigational Site Number 0324002, Caba
  - Investigational Site Number 0324005, Ciudad Autónoma Buenos Aires
  - Investigational Site Number 0324008, Córdoba
  - Investigational Site Number 0324006, Córdoba
  - Investigational Site Number 0324009, La Plata
  - Investigational Site Number 0324007, Mar del Plata
- Brazil (7):
  - Investigational Site Number 0764001, Belém
  - Investigational Site Number 0764007, Belo Horizonte
  - Investigational Site Number 0764002, Curitiba
  - Investigational Site Number 0764008, Curitiba
  - Investigational Site Number 0764005, Rio de Janeiro
  - Investigational Site Number 0764004, São Paulo
  - Investigational Site Number 0764006, São Paulo
- Canada (10):
  - Investigational Site Number 1244007, Brampton
  - Investigational Site Number 1244004, Burlington
  - Investigational Site Number 1244005, Etobicoke
  - Investigational Site Number 1244006, Laval
  - Investigational Site Number 1244009, Montreal
  - Investigational Site Number 1244010, Ottawa
  - Investigational Site Number 1244003, Thornhill
  - Investigational Site Number 1244002, Toronto
  - Investigational Site Number 1244008, Toronto
  - Investigational Site Number 1244001, Vancouver
- Colombia (8):
  - Investigational Site Number 1704008, Barranquilla
  - Investigational Site Number 1704007, Barranquilla
  - Investigational Site Number 1704004, Bogotá
  - Investigational Site Number 1704009, Bogotá
  - Investigational Site Number 1704006, Ibagué
  - Investigational Site Number 1704001, Manizales
  - Investigational Site Number 1704002, Medellin / Antioquia
  - Investigational Site Number 1704005, Zipaquirá
- Germany (3):
  - Investigational Site Number 2764001, Frankfurt am Main
  - Investigational Site Number 2764002, Hamburg
  - Investigational Site Number 2764003, Münster
- Hungary (10):
  - Investigational Site Number 3484008, Baja
  - Investigational Site Number 3484012, Baja
  - Investigational Site Number 3484002, Balatonfüred
  - Investigational Site Number 3484007, Budapest
  - Investigational Site Number 3484011, Debrecen
  - Investigational Site Number 3484005, Debrecen
  - Investigational Site Number 3484001, Gyula
  - Investigational Site Number 3484010, Nyíregyháza
  - Investigational Site Number 3484013, Nyregyhza
  - Investigational Site Number 3484004, Pécs
- Israel (12):
  - Investigational Site Number 3764001, Ashkelon
  - Investigational Site Number 3764010, Beersheba
  - Investigational Site Number 3764007, Haifa
  - Investigational Site Number 3764009, Kfar Saba
  - Investigational Site Number 3764011, Kfar Saba
  - Investigational Site Number 3764003, Nahariya
  - Investigational Site Number 3764004, Petah Tikva
  - Investigational Site Number 3764006, Ramat Gan
  - Investigational Site Number 3764005, Rehovot
  - Investigational Site Number 3764008, Safed
  - Investigational Site Number 3764002, Tel Aviv
  - Investigational Site Number 3764013, Ẕerifin
- Italy (7):
  - Investigational Site Number 3804007, Catania
  - Investigational Site Number 3804005, Milan
  - Investigational Site Number 3804004, Milan
  - Investigational Site Number 3804008, Naples
  - Investigational Site Number 3804002, Napoli
  - Investigational Site Number 3804003, Roma
  - Investigational Site Number 3804006, Siena
- Mexico (7):
  - Investigational Site Number 4844009, Chihuahua Chihuahua
  - Investigational Site Number 4844008, Durango, Durango
  - Investigational Site Number 4844001, Guadalajara
  - Investigational Site Number 4844003, Guadalajara
  - Investigational Site Number 4844006, Merida, Yucatan
  - Investigational Site Number 4844005, Monterrey
  - Investigational Site Number 4844004, Xalapa
- Poland (11):
  - Investigational Site Number 6164002, Bialystok
  - Investigational Site Number 6164006, Katowice
  - Investigational Site Number 6164010, Krakow
  - Investigational Site Number 6164009, Krakow
  - Investigational Site Number 6164004, Krakow
  - Investigational Site Number 6164008, Krakow
  - Investigational Site Number 6164011, Lodz
  - Investigational Site Number 6164005, Oświęcim
  - Investigational Site Number 6164003, Rzeszów
  - Investigational Site Number 6164012, Skierniewice
  - Investigational Site Number 6164007, Warsaw
- Romania (8):
  - Investigational Site Number 6424002, Bacau
  - Investigational Site Number 6424001, Bacau
  - Investigational Site Number 6424004, Bucharest
  - Investigational Site Number 6424009, Bucharest
  - Investigational Site Number 6424010, Bucharest
  - Investigational Site Number 6424006, Hunedoara
  - Investigational Site Number 6424011, Oradea
  - Investigational Site Number 6424003, Târgu Mureş
- Russia (6):
  - Investigational Site Number 6434003, Chelyabinsk
  - Investigational Site Number 6434005, Kemerovo
  - Investigational Site Number 6434002, Krasnodar
  - Investigational Site Number 6434004, Novosibirsk
  - Investigational Site Number 6434001, Saint Petersburg
  - Investigational Site Number 6434006, Yaroslavl
- South Africa (6):
  - Investigational Site Number 7104008, Cape Town
  - Investigational Site Number 7104002, Cape Town
  - Investigational Site Number 7104001, Johannesburg
  - Investigational Site Number 7104010, Johannesburg
  - Investigational Site Number 7104005, Johannesburg
  - Investigational Site Number 7104006, Pretoria
- Spain (7):
  - Investigational Site Number 7244011, Barcelona
  - Investigational Site Number 7244007, Granada
  - Investigational Site Number 7244003, Madrid
  - Investigational Site Number 7244006, Palma de Mallorca
  - Investigational Site Number 7244001, Seville
  - Investigational Site Number 7244002, Valencia
  - Investigational Site Number 7244009, Zaragoza
- Ukraine (10):
  - Investigational Site Number 8044004, Dnipropetrovsk
  - Investigational Site Number 8044007, Kharkiv
  - Investigational Site Number 8044010, Kharkiv
  - Investigational Site Number 8044008, Kiev
  - Investigational Site Number 8044003, Kiev
  - Investigational Site Number 8044009, Kyiv
  - Investigational Site Number 8044001, Kyiv
  - Investigational Site Number 8044006, Kyiv
  - Investigational Site Number 8044005, Lviv
  - Investigational Site Number 8044002, Zaporizhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cherney DZI, Ferrannini E, Umpierrez GE, Peters AL, Rosenstock J, Powell DR, Davies MJ, Banks P, Agarwal R. Efficacy and safety of sotagliflozin in patients with type 2 diabetes and stage 3 chronic kidney disease. Diabetes Obes Metab. 2023 Jun;25(6):1646-1657. doi: 10.1111/dom.15019. Epub 2023 Feb 28. PMID 36782093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 166 investigative sites in the United States, Argentina, Brazil, Canada, Colombia, Germany, Hungary, Israel, Italy, Mexico, Poland, Romania, Russian Federation, South Africa, Spain, and Ukraine from 16 August 2017 to 25 October 2019.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus were enrolled in 1 of 3 treatment groups: Placebo or Sotagliflozin 200 milligrams (mg) or Sotagliflozin 400 mg. Participants were randomly assigned in the ratio of 1:1:1 to these reporting groups.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 260 | 263 | 264
Completed | 224 | 240 | 232
Not Completed | 36 | 23 | 32
Not completed — At the Participant's own Request | 18 | 10 | 15
Not completed — Adverse Event | 8 | 6 | 9
Not completed — Poor Compliance to Protocol | 0 | 2 | 3
Not completed — Study Terminated by Sponsor | 1 | 0 | 0
Not completed — Reason not Specified | 4 | 4 | 1
Not completed — Lost to Follow-up | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants or participants analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 260 | 263 | 264 | 787
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (8.1) | 69.6 (7.5) | 69.5 (8.2) | 69.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 120 | 112 | 343
  Male | 149 | 143 | 152 | 444
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 67 | 64 | 198
  Not Hispanic or Latino | 193 | 196 | 200 | 589
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 9 | 20 | 44
  Asian | 5 | 7 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 12 | 14 | 15 | 41
  White | 220 | 231 | 215 | 666
  More than one race | 3 | 0 | 3 | 6
  Unknown or Not Reported | 4 | 1 | 3 | 8
Region of Enrollment [Number; unit: participants]
  Colombia | 12 | 6 | 14 | 32
  Argentina | 8 | 8 | 8 | 24
  Romania | 6 | 14 | 13 | 33
  Hungary | 21 | 23 | 13 | 57
  United States | 66 | 72 | 62 | 200
  Ukraine | 12 | 13 | 14 | 39
  Spain | 9 | 10 | 15 | 34
  Russia | 15 | 10 | 14 | 39
  Canada | 11 | 18 | 12 | 41
  Poland | 29 | 23 | 32 | 84
  Brazil | 22 | 22 | 22 | 66
  Italy | 5 | 6 | 8 | 19
  South Africa | 7 | 3 | 12 | 22
  Mexico | 14 | 13 | 7 | 34
  Israel | 23 | 17 | 16 | 56
  Germany | 0 | 5 | 2 | 7
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] — Population: Number analyzed specifies the number of participants evaluated for the parameter.
  percentage of HbA1c
    number analyzed (Participants) | 260 | 262 | 264 | 786
    (all) | 8.33 (1.00) | 8.33 (0.9) | 8.31 (0.94) | 8.32 (0.95)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 140.59 (14.59) | 140.31 (15.15) | 141.71 (15.01) | 140.87 (14.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 26
Description: An Analysis of covariance (ANCOVA) model was used for analysis.
Time Frame: Baseline to Week 26
Population: Intent-to-treat (ITT) population included all randomized participants or participants analyzed according to their randomized treatment. Missing data was imputed using control-based copy reference multiple imputation under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 263 | 264
percentage of HbA1c | -0.22 (0.061) | -0.32 (0.060) | -0.46 (0.060)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, randomization stratum of Chronic Kidney Disease (CKD) stage (3A, 3B) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p = 0.2095, ANCOVA; Difference in Least Squares (LS) Means = -0.1, 95% CI 2-sided [-0.245 to 0.054], Standard Error of Mean 0.076
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, randomization stratum of CKD stage (3A, 3B) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p = 0.0021, ANCOVA; Difference in LS Means = -0.24, 95% CI 2-sided [-0.386 to -0.085], Standard Error of Mean 0.077

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: An ANCOVA model was used for analysis.
Time Frame: Baseline to Week 26
Population: ITT population included all randomized participants or participants analyzed according to their randomized treatment. Missing data was imputed using the retrieved dropouts & washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 263 | 264
millimole per liter (mmol/L) | -0.374 (0.1949) | -0.961 (0.1715) | -0.852 (0.1668)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, randomization stratum of CKD stage (3A, 3B) at screening, and country as fixed effects, and baseline FPG as a covariate; Test type: Superiority; p = 0.0144, ANCOVA; Difference in LS Means = -0.587, 95% CI 2-sided [-1.0564 to -0.1169], Standard Error of Mean 0.2397
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0436, ANCOVA; Difference in LS Means = -0.478, 95% CI 2-sided [-0.942 to -0.0136], Standard Error of Mean 0.2368

3. Secondary Outcome: Change From Baseline in SBP for Participants With Baseline SBP ≥130 mmHg at Week 12
Description: An ANCOVA model was used for analysis.
Time Frame: Baseline to Week 12
Population: Analysis population included participants with baseline SBP ≥130 mmHg in ITT population where, ITT population included all randomized participants or participants analyzed according to their randomized treatment. Missing data was imputed using the retrieved dropouts & washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 175 | 162 | 182
mmHg | -5.18 (1.462) | -7.46 (1.597) | -7.71 (1.247)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 12 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization stratum of CKD stage (3A, 3B) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.2627, ANCOVA; Difference in LS Means = -2.28, 95% CI 2-sided [-6.265 to 1.709], Standard Error of Mean 2.034
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1602, ANCOVA; Difference in LS Means = -2.53, 95% CI 2-sided [-6.052 to 1], Standard Error of Mean 1.799

4. Secondary Outcome: Change From Baseline in SBP at Week 12 for All Participants
Description: An ANCOVA model was used for analysis.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 263 | 264
mmHg | -3.31 (1.037) | -4.91 (1.010) | -4.94 (0.983)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 12 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, randomization stratum of CKD stage (3A, 3B) at screening, country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.2212, ANCOVA; Difference in LS Means = -1.59, 95% CI 2-sided [-4.142 to 0.958], Standard Error of Mean 1.301
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.2089, ANCOVA; Difference in LS Means = -1.63, 95% CI 2-sided [-4.171 to 0.912], Standard Error of Mean 1.297

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: An ANCOVA model was used for analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 263 | 264
kilogram (kg) | -0.38 (0.262) | -1.66 (0.246) | -1.20 (0.257)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, randomization stratum of CKD stage (3A, 3B) at screening, country as fixed effects, and baseline body weight as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.28, 95% CI 2-sided [-1.92 to -0.644], Standard Error of Mean 0.326
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0155, ANCOVA; Difference in LS Means = -0.82, 95% CI 2-sided [-1.487 to -0.156], Standard Error of Mean 0.339

6. Secondary Outcome: Percentage Change From Baseline in the Urine Albumin: Creatinine Ratio (UACR) at Week 26 in Participants With Baseline UACR >30 Milligrams Per Gram (mg/g)
Description: An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated.
Time Frame: Baseline to Week 26
Population: Analysis population included participants with baseline UACR >30 mg/g in ITT population where, ITT population included all randomized participants or participants analyzed according to their randomized treatment. Missing data was imputed using control-based copy reference multiple imputation under the missing not at random framework.
Measure: Geometric Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 263 | 264
percent change | -18.71 (NA) — An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated. | -43.68 (NA) — An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated. | -48.12 (NA) — An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated.
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, randomization stratum of CKD stage (3A, 3B) at screening, country as fixed effects, and and log-transformed baseline UACR as a covariate; Test type: Superiority; p = 0.0015, ANCOVA; Percent Difference = -30.72, 95% CI 2-sided [-44.78 to -13.07]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA; Percent Difference = -36.18, 95% CI 2-sided [-49.91 to -18.68]

7. Secondary Outcome: Percentage of Participants With HbA1c <6.5% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants or participants analyzed according to their randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 263 | 264
percentage of participants | 4.2 | 5.7 | 5.7
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Percentage difference between treatment groups using the Cochran-Mantel-Haenszel test stratified by the randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening and randomization strata of CKD stage (3A, 3B) at screening; Test type: Superiority; p = 0.4328, Cochran-Mantel-Haenszel; Percentage Difference = 1.5, 95% CI 2-sided [-2.23 to 5.21]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.4328, Cochran-Mantel-Haenszel; Percentage Difference = 1.5, 95% CI 2-sided [-2.2 to 5.17]

8. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants or participants analyzed according to their randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 263 | 264
percentage of participants | 13.5 | 19.4 | 20.8
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0614, Cochran-Mantel-Haenszel; Percentage Difference = 6, 95% CI 2-sided [-0.23 to 12.21]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel; Percentage Difference = 7.4, 95% CI 2-sided [1.08 to 13.65]

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Up to 60 weeks
Population: Safety population included all participants who received at least 1 dose of study drug analyzed according to the treatment actually received.
Measure: Number; unit: percentage of participants
Groups:
- Sotagliflozin 200 mg: Following a 2-week run-in period, participants received two tablets, 1 sotagliflozin 200 mg tablet and 1 placebo tablet (identical to sotagliflozin 200 mg in appearance), orally once daily, before the first meal of the day for up to 58 weeks. Four participants randomized to sotagliflozin 400 mg were dosed with both sotagliflozin 200 mg and 400 mg. These participants were included in the sotagliflozin 200 mg arm in the safety population.
- Sotagliflozin 400 mg: Following a 2-week run-in period, participants received sotagliflozin 400 mg, administered as two 200 mg sotagliflozin tablets, orally once daily, before the first meal of the day for up to 60 weeks. Four participants randomized to sotagliflozin 400 mg were dosed with both sotagliflozin 200 mg and 400 mg. These participants were included in the sotagliflozin 200 mg arm in the safety population.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 267 | 260
percentage of participants | 78.1 | 76.8 | 74.2

10. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events
Description: Percentage of participants with hypoglycemic events are reported for the following 3 categories: Any hypoglycemia (as reported in the Electronic Case Report Form); Documented symptomatic hypoglycemia [typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤ 70 mg/dL (3.9 mmol/L)]; Severe [an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions] or documented symptomatic hypoglycemia [typical symptoms of hypoglycemia and plasma glucose ≤ 70 mg/dL].
Time Frame: Up to 60 weeks
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Following a 2-week run-in phase, participants received two placebo tablets (identical to Sotagliflozin 200 mg in appearance), orally once daily for up to 54 weeks.
- Sotagliflozin 200 mg: Following a 2-week run-in phase, participants received two tablets, 1 Sotagliflozin 200 mg tablet and 1 placebo tablet (identical to Sotagliflozin 200 mg in appearance), orally once daily for up to 58 weeks. Four participants randomized to Sotagliflozin 400 mg were dosed with both Sotagliflozin 200 mg and 400 mg. These participants were included in the Sotagliflozin 200 mg arm in the safety population.
- Sotagliflozin 400 mg: Following a 2-week run-in phase, participants received Sotagliflozin 400 mg, administered as two 200 mg Sotagliflozin tablets, orally once daily for up to 60 weeks. Four participants randomized to Sotagliflozin 400 mg were dosed with both Sotagliflozin 200 mg and 400 mg. These participants were included in the Sotagliflozin 200 mg arm in the safety population.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 260 | 267 | 260
percentage of participants
  Any hypoglycemia | 38.1 | 41.9 | 35.4
  Documented symptomatic hypoglycemia | 26.9 | 29.6 | 22.3
  Severe or documented symptomatic hypoglycemia | 26.9 | 29.6 | 22.3

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Description: Safety population included all participants who received at least 1 dose of study drug analyzed according to the treatment actually received. Four participants randomized to sotagliflozin 400 mg were dosed with both sotagliflozin 200 mg and 400 mg. These participants were included in the sotagliflozin 200 mg arm in the safety population. Hypoglycemia was captured and handled separately from other adverse events and is reported in the outcome measure section.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 3/260 | 2/267 | 5/260
Serious Adverse Events (participants affected / at risk) | 48/260 | 43/267 | 44/260
Other Adverse Events (participants affected / at risk) | 80/260 | 72/267 | 77/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=260) | Sotagliflozin 200 mg (N=267) | Sotagliflozin 400 mg (N=260)
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 2 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac death (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural shock (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 2
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 4 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 3 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 2 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 0
Iris neovascularisation (Eye disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 2
End stage renal disease (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Corneal abscess (Infections and infestations) | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 1 | 0
Funguria (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 2 | 0 | 0
Infective periostitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1
Sepsis pasteurella (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Tick-borne viral encephalitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=260) | Sotagliflozin 200 mg (N=267) | Sotagliflozin 400 mg (N=260)
Diarrhoea (Gastrointestinal disorders) | 13 | 15 | 22
Vitamin D deficiency (Metabolism and nutrition disorders) | 30 | 24 | 24
Nasopharyngitis (Infections and infestations) | 13 | 7 | 12
Upper respiratory tract infection (Infections and infestations) | 18 | 16 | 13
Urinary tract infection (Infections and infestations) | 21 | 19 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT03242252/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03242252/SAP_001.pdf